CLINICAL TRIAL: NCT04854434
Title: A Phase 2 Open-Label Multicenter Study to Evaluate the Safety and Efficacy of Selinexor With or Without Pembrolizumab Versus Standard of Care in Previously Treated Metastatic Colorectal Cancer With RAS Mutations
Brief Title: A Study to Evaluate the Safety and Efficacy of Selinexor With or Without Pembrolizumab Versus Standard of Care in Previously Treated Metastatic Colorectal Cancer With RAS Mutations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XPORT-CRC-041
Record Dates: First submitted 2021-04-17; First posted 2021-04-22 (Actual); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — selinexor; pembrolizumab; Trifluridine; tipiracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Selinexor 80 mg (Experimental): Participants received a single dose of selinexor 80 mg (4 tablets of 20 mg) orally QW on Day 1 of each week of a 42-day cycle (i.e., on Days 1, 8, 15, 22, 29, and 36 of each 42-day cycle) until PD, intolerable toxicity, or withdrawal from the study (maximum exposure: 33 weeks).
  Interventions: Drug: Selinexor
- Arm B: Selinexor 80 mg and Pembrolizumab 400 mg (Experimental): Participants received a single dose of selinexor 80 mg (4 tablets of 20 mg) orally QW on Day 1 of each week of a 42-day cycle (i.e., on Days 1, 8, 15, 22, 29, and 36 of each 42-day cycle) in combination with pembrolizumab 400 mg IV once every 6 weeks of each 42-day cycle until PD, intolerable toxicity, or withdrawal from the study (maximum exposure: 30 weeks).
  Interventions: Drug: Selinexor; Drug: Pembrolizumab
- Arm C: Standard of care (SOC) (Active Comparator): Participants received combination of trifluridine and tipiracil 35 mg/m^2/dose tablets orally BID (maximum 80 mg per dose) as SOC on Days 1 through 5 and Days 8 through 12 of each 28-day cycle until PD, intolerable toxicity, or withdrawal from the study (maximum exposure: 11 weeks).
  Interventions: Drug: Trifluridine; Drug: Tipiracil

INTERVENTIONS:
Drug: Selinexor — Participants will receive selinexor oral tablets.
  Other Names: Xpovio; KPT-330
  Arms: Arm A: Selinexor 80 mg; Arm B: Selinexor 80 mg and Pembrolizumab 400 mg
Drug: Pembrolizumab — Participants will receive pembrolizumab intravenously.
  Other Names: Keytruda
  Arms: Arm B: Selinexor 80 mg and Pembrolizumab 400 mg
Drug: Trifluridine — Participants will receive trifluridine oral tablets as SOC.
  Arms: Arm C: Standard of care (SOC)
Drug: Tipiracil — Participants will receive tipiracil oral tablets as SOC.
  Arms: Arm C: Standard of care (SOC)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of selinexor alone or with pembrolizumab in participants with advanced or metastatic colorectal cancer (CRC). Approximately 78 participants with advanced or metastatic CRC will be enrolled, and randomized (1:1:1) into three arms A (selinexor only), B (selinexor and pembrolizumab), and C (standard of care [Combination of trifluridine and tipiracil]). Randomization will be based on stratification factors: Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 versus 2. The end of treatment (EoT) visit will occur less than or equal to (<=30) days post-treatment discontinuation. A survival follow-up visit will be performed every 3 months from EoT and will continue for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants have histologically proven diagnosis of unresectable metastatic colorectal cancer with a known rat sarcoma (RAS) mutation.
* Participants have measurable disease according to RECIST 1.1 criteria.
* Have received 2-3 prior lines of systemic anticancer treatment (adjuvant or neoadjuvant therapy is not counted as one line of systemic therapy).
* Participants with stable previously treated brain metastases are allowed.
* ECOG performance status of 0-2 at the time of screening.
* Age ≥ 18 years at the time of signing informed consent
* Life expectancy of at least 3 months.
* Female participants of childbearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male participants must use an effective barrier method of contraception if sexually active throughout the study and for 4 months after the last dose of selinexor or pembrolizumab or 6 months after trifluridine and tipiracil.
* Written informed consent signed in accordance with federal, local, and institutional guidelines.

Exclusion Criteria:

* Prior treatment with a selective inhibitor of nuclear export (SINE) compound or selinexor.
* Prior treatment with immune checkpoint inhibitors.
* Participants with microsatellite instability high (MSI-H) or deficient mismatch repair (dMMR).
* Known allergy to any of study drugs (selinexor, pembrolizumab, and trifluridine and tipiracil) or the excipient of pembrolizumab.
* Significant cardiovascular impairment, defined as:

  * Left ventricular ejection fraction ≤ 40 percent (%)
  * Active congestive heart failure (New York Heart Association [NYHA]) Class ≥ 3
  * Unstable angina or myocardial infarction within 3 months of enrollment
  * Serious and potentially life-threatening arrhythmia
* Impaired hematopoietic function (any of the following would result in exclusion):

  * Absolute neutrophil count (ANC) less than (<) 1500/cubic millimeter (mm^3)
  * Platelet count < 100,000/ mm^3
  * Hemoglobin (Hb) < 10 gram per deciliter (g/dL)
* Significant renal impairment, defined as: calculated creatinine clearance (CrCl) of < 30 milliliter per minute (mL/min) using the formula of Cockcroft and Gault.
* Impaired hepatic function defined as: total bilirubin greater than (>) 1.5 × upper limit of normal (ULN) and aspartate transaminase (AST) > 2.5 x ULN, AST > 2.5 x ULN; for Arm B, unless bilirubin elevation is related to Gilbert's Syndrome for which bilirubin must be ≤ 4 x ULN.
* Participants with a diagnosis of immunodeficiency or are receiving systemic steroid therapy (>10 mg/day of prednisone or equivalent) or any other form of immunosuppressive therapy. Participants with active autoimmune disease requiring systemic treatment during the past 2 years.

  * Participants with controlled type I and type II diabetes mellitus, and endocrinopathies such as hypothyroidism on stable hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are allowed.

Note: The Investigator needs to evaluate the participants medical history to confirm that they are eligible to receive the combination with pembrolizumab per these criteria.

* Insufficient time since or not recovered from procedures or anti-cancer therapy, defined as:

  * Not recovered from major surgery ≤ 21 days prior to Day 1 dosing. Minor procedures, such as biopsies, dental work, or placement of a port or IV line for infusion are permitted.
  * Have ongoing clinically significant anti-cancer therapy-related toxicities Common Terminology Criteria for Adverse Events (CTCAE) Grade > 1. In specific cases, participants whose toxicity has stabilized or with Grade 2 non-hematologic toxicities can be allowed following documented approval by the Sponsor's Medical Monitor.
  * Had last dose of previous anti-cancer therapy ≤14 days prior to Day 1 dosing.
  * Palliative radiotherapy > 14 days prior to the study is allowed.
  * Received investigational drugs in other clinical trials within 28 days, or 5 half-lives of the investigational drug (whichever is shorter), prior to Cycle 1 Day 1 (C1D1).
  * Live-attenuated vaccine against an infectious disease (e.g., nasal spray influenza vaccine) ≤ 14 days prior to the intended C1D1.
* Female participants who are pregnant or lactating.
* Active, ongoing or uncontrolled active infection requiring parenteral antibiotics, antivirals, antifungals within 1 week of Screening.
* Participants with autoimmune disease, a medical condition that requires systemic corticosteroids or other immunosuppressive medication; or a history of interstitial lung disease.
* Any gastrointestinal dysfunctions that could interfere with the absorption of selinexor (e.g. bowel obstruction, inability to swallow tablets, malabsorption syndrome, unresolved nausea, vomiting, diarrhea CTCAE > grade 1).
* In the opinion of the investigator, participants who are below their ideal body weight and would be unduly impacted by changes in their weight.
* Serious psychiatric or medical conditions that could interfere with participation in the study or in the opinion of the Investigator would make study involvement unreasonably hazardous.
* Concurrent therapy with approved or investigational anticancer therapeutic including topical therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Christiana Care Health Services, Christiana Hospital, Newark, Delaware
  - BRCR Global, Plantation, Florida

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 investigational sites in the United States.
Pre-assignment Details: A total of 13 participants were enrolled and randomized to receive study treatments Arm A (single-agent selinexor), Arm B (selinexor + pembrolizumab), or Arm C (standard of care) based on the stratification factor of Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 versus 2.
Groups:
- Arm A: Selinexor 80 mg: Participants received a single dose of selinexor 80 milligrams (mg); (4 tablets of 20 mg) orally once weekly (QW) on Day 1 of each week of a 42-day cycle (i.e., on Days 1, 8, 15, 22, 29, and 36 of each 42-day cycle) until progressive disease (PD), intolerable toxicity, or withdrawal from the study (maximum exposure: 33 weeks).
- Arm B: Selinexor 80 mg and Pembrolizumab 400 mg: Participants received a single dose of selinexor 80 mg (4 tablets of 20 mg) orally QW on Day 1 of each week of a 42-day cycle (i.e., on Days 1, 8, 15, 22, 29, and 36 of each 42-day cycle) in combination with pembrolizumab 400 mg intravenously (IV) once every 6 weeks of each 42-day cycle until PD, intolerable toxicity, or withdrawal from the study (maximum exposure: 30 weeks).
- Arm C: Standard of Care (SOC): Participants received combination of trifluridine and tipiracil 35 milligrams per square meter per dose (mg/m^2/dose) tablets orally twice daily (BID) (maximum 80 mg per dose) as SOC on Days 1 through 5 and Days 8 through 12 of each 28-day cycle until PD, intolerable toxicity, or withdrawal from the study (maximum exposure: 11 weeks).
Period: Overall Study
Arm/Group | Arm A: Selinexor 80 mg | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC)
Started | 4 | 5 | 4
Completed | 0 | 1 | 0
Not Completed | 4 | 4 | 4
Not completed — Death | 1 | 3 | 4
Not completed — Study Terminated by Sponsor | 2 | 0 | 0
Not completed — Other | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Selinexor 80 mg | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC) | Total
Number analyzed (Participants) | 4 | 5 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (3.11) | 61.0 (14.78) | 57.0 (17.63) | 62.7 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 1 | 6
  Male | 3 | 1 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 3 | 5 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 3 | 5 | 4 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Arm B and C: Progression-free Survival (PFS) as Assessed by the Investigator Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: PFS was defined as the time from the date of randomization until disease progression or death due to any cause, whichever occurs first. PFS was assessed by the investigator per RECIST 1.1. As per RECIST 1.1 criteria, PD was defined as at least a 20% increase in the sum of the longest diameter (SLD), taking as reference the smallest sum of the longest diameter (SLD) recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From the date of randomization until disease progression or death, whichever occurs first (up to 8 months)
Population: Prior to study completion, the signal was assessed by sponsor to be uncompetitive in the current treatment landscape and thus the colorectal cancer (CRC) program was closed. Data for this outcome measure was not planned to be collected and analyzed for Arm A.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 5 | 4
Months | NA [NA to NA] — Median PFS and 95% CI was not available due to insufficient numbers of participants with events. | NA [NA to NA] — Median PFS and 95% CI was not available due to insufficient numbers of participants with events.

2. Secondary Outcome: Arm A, B and C: Overall Survival (OS)
Description: OS was defined as time from the date of randomization to death due to any cause.
Time Frame: From the date of randomization up to death (up to 8 months)
Population: Prior to study completion, the signal was assessed by sponsor to be uncompetitive in the current treatment landscape and thus CRC program was closed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Selinexor 80 mg | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 4 | 5 | 4
months | NA [NA to NA] — Median and 95% CI was not available due to insufficient numbers of participants with events. | NA [NA to NA] — Median and 95% CI was not available due to insufficient numbers of participants with events. | NA [NA to NA] — Median and 95% CI was not available due to insufficient numbers of participants with events.

3. Secondary Outcome: Arm B and C: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieve complete response (CR) or partial response (PR) or or initiating a new antineoplastic therapy. ORR was assessed by RECIST 1.1 as defined by the Investigator based on radiologic criteria. Per RECIST 1.1 criteria, CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization until the documentation of CR or PR, whichever occurs first (up to 8 months)
Population: ITT population included all participants randomized to study treatment and were analyzed in the treatment arm to which they were randomized. Data for this outcome measure was not planned to be collected and analyzed for Arm A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 5 | 4
percentage of participants | 0 [NA to NA] — Lower limit and upper limit of 95% confidence interval was not available because no participant had CR/PR event. | 0 [NA to NA] — Lower limit and upper limit of 95% confidence interval was not available because no participant had CR/PR event.

4. Secondary Outcome: Arm A and C: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieve CR or PR or or initiating a new antineoplastic therapy. ORR was assessed by RECIST 1.1 as defined by the Investigator based on radiologic criteria. Per RECIST 1.1 criteria, CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization until the documentation of CR or PR, whichever occurs first (up to 8 months)
Population: ITT population included all participants randomized to study treatment and were analyzed in the treatment arm to which they were randomized. Data for this outcome measure was not planned to be collected and analyzed for Arm B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Selinexor 80 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 4 | 4
percentage of participants | 25.0 [0.6 to 80.6] | 0 [NA to NA] — Lower limit and upper limit of 95% confidence interval was not available because no participant had CR/PR event.

5. Secondary Outcome: Arm A, B and C: Progression-free Survival (PFS) at 6 Months
Description: PFS at 6 months was defined as the time from the date of randomization without disease progression at 6 months as assessed by the investigator per RECIST 1.1. As per RECIST 1.1 criteria, PD was defined as at least a 20% increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: At 6 Months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Selinexor 80 mg | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 4 | 5 | 4
months | NA [NA to NA] — Median PFS and 95% CI was not available due to insufficient numbers of participants with events. | NA [NA to NA] — Median PFS and 95% CI was not available due to insufficient numbers of participants with events. | NA [NA to NA] — Median PFS and 95% CI was not available due to insufficient numbers of participants with events.

6. Secondary Outcome: Arm A, B and C: Percentage of Participants With Overall Survival (OS) at 6 Months
Description: OS was defined as the time from the first dose date to date of death due to any cause. Participant was considered as event (overall survival) free if participant was not died and was alive at 6 months.
Time Frame: At 6 Months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: percentage of event free participants
Arm/Group | Arm A: Selinexor 80 mg | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 4 | 5 | 4
percentage of event free participants | NA [NA to NA] — Median and 95% CI was not available due to insufficient numbers of participants with events. | NA [NA to NA] — Median and 95% CI was not available due to insufficient numbers of participants with events. | NA [NA to NA] — Median and 95% CI was not available due to insufficient numbers of participants with events.

7. Secondary Outcome: Arm A, B and C: Percentage of Participants With Overall Survival (OS) at 12 Months
Description: OS was defined as the time from the first dose date to date of death due to any cause. Participant was considered as event (overall survival) free if participant was not died and was alive at 12 months.
Time Frame: At 12 Months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: percentage of event free participants
Arm/Group | Arm A: Selinexor 80 mg | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 4 | 5 | 4
percentage of event free participants | NA [NA to NA] — Median and 95% CI was not available due to insufficient numbers of participants with events. | NA [NA to NA] — Median and 95% CI was not available due to insufficient numbers of participants with events. | NA [NA to NA] — Median and 95% CI was not available due to insufficient numbers of participants with events.

8. Secondary Outcome: Arm B and C: Duration of Response (DOR) Based on Response Evaluation Criteria in Solid Tumors Version 1.1
Description: DOR was defined as the time from first occurrence of CR or PR until the first date of PD per RECIST version 1.1 or death. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first occurrence of CR or PR until disease progression or death, whichever occurs first (up to 8 months)
Population: ITT population included all participants randomized to study treatment and were analyzed in the treatment arm to which they were randomized. Here, "overall number of participants analyzed" signifies those who had response (CR/PR) in specified arm. Data for this outcome measure was not planned to be collected and analyzed for Arm A.
Arm/Group | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Arm A and C: Duration of Response (DOR) Based on Response Evaluation Criteria in Solid Tumors Version 1.1
Description: as for outcome 8
Time Frame: From first occurrence of CR or PR until disease progression or death, whichever occurs first (up to 8 months)
Population: ITT population included all participants randomized to study treatment and were analyzed in the treatment arm to which they were randomized. Here, "overall number of participants analyzed" signifies those who had response (CR/PR) in specified arm. Data for this outcome measure was not planned to be collected and analyzed for Arm B.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Selinexor 80 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 1 | 0
months | NA [NA to NA] — Median and 95% CI was not estimable due to single participant. |

10. Secondary Outcome: Arm B and C: Percentage of Participants With Confirmed Disease Control Rate as Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: Disease control rate was defined as participants who achieved best overall response of CR, PR, or at least 12 continuous weeks of stable disease (SD) as assessed by investigator as per RECIST v 1.1. As per RECIST v 1.1 before PD or initiating a new antineoplastic therapy, CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (at least a 20% increase in the sum of diameters of target lesions) taking as reference the smallest sum diameters while on study.
Time Frame: From the date of randomization up to death (up to 8 months)
Population: ITT population included all participants randomized to study treatment and were analyzed in the treatment arm to which they were randomized. Here, "overall number of participants analyzed" signifies those who had response (CR/PR/SD) in specified arm. Data for this outcome measure was not planned to be collected and analyzed for Arm A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 5 | 0
percentage of participants | 40.0 [5.3 to 85.3] |

11. Secondary Outcome: Arm A and C: Percentage of Participants With Confirmed Disease Control Rate as Per Response Evaluation Criteria in Solid Tumors Version 1.1
Description: as for outcome 10
Time Frame: From the date of randomization up to death (up to 8 months)
Population: ITT population included all participants randomized to study treatment and were analyzed in the treatment arm to which they were randomized. Here, "overall number of participants analyzed" signifies those who had response (CR/PR/SD) in specified arm. Data for this outcome measure was not planned to be collected and analyzed for Arm B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Selinexor 80 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 4 | 0
percentage of participants | 100 [NA to NA] — Lower limit and upper limit of 95% confidence interval was not available because all participants had CR/PR/SD event. |

12. Secondary Outcome: Arm A, B and C: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. A SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. A TEAE was defined as those AEs that develop or worsen after the first dose of study drug. TEAEs included both serious and non-serious TEAEs.
Time Frame: From start of study drug administration up to 12 months
Population: Safety population included all participants who were assigned to study treatment and who received greater than or equal to 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Selinexor 80 mg | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC)
Number analyzed (Participants) | 4 | 5 | 4
Participants
  Participants with TEAEs | 4 | 5 | 4
  Participants with Serious TEAEs | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 12 months
Description: Analysis was performed on safety population.
Arm/Group | Arm A: Selinexor 80 mg | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg | Arm C: Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 1/4 | 3/5 | 4/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/5 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Selinexor 80 mg (N=4) | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg (N=5) | Arm C: Standard of Care (SOC) (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Selinexor 80 mg (N=4) | Arm B: Selinexor 80 mg and Pembrolizumab 400 mg (N=5) | Arm C: Standard of Care (SOC) (N=4)
Nausea (Gastrointestinal disorders) | 3 | 4 | 3
Fatigue (General disorders) | 1 | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Asthenia (General disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Androgen deficiency (Endocrine disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Temperature intolerance (General disorders) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Protein total decreased (Investigations) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Prior to study completion, the signal was assessed by sponsor to be uncompetitive in the current treatment landscape and thus CRC program was closed. Thereby some of the protocol planned analysis were not performed and thus no data was reported for those outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT04854434/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT04854434/SAP_001.pdf